CLINICAL TRIAL: NCT05592327
Title: Citric Acid Passivation on Implant Abutments for the Prevention of Peri-implant Disease: a Randomized Controlled Clinical Trial
Brief Title: Citric Acid Passivation on Implant Abutments for the Prevention of Peri-implant Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Klockner Implant System (Unknown)
Responsible Party: Principal Investigator, Javi Vilarrasa, Doctor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PER-ECL-2021-04
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Peri-Implantitis; Implant Infection; Microbial Disease
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, triple blind, controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citric acid abutment (Experimental): Antimicrobial-coated abutments (citric acid) will be allocated to the test group.
  Permanent Vega® (Klockner Implant System, Barcelona, Spain) will be used. The interface between implant and abutment is platform switching. The abutment height will be of 2 mm. It will be placed the day of the implant surgery and tighten to 25 N
  Interventions: Procedure: Citric acid abutment
- Control non coated abutment (Placebo Comparator): Non- coated abutments (citric acid) will be allocated to the control group. Permanent Vega® (Klockner Implant System, Barcelona, Spain) will be used. The interface between implant and abutment is platform switching. The abutment height will be of 2 mm. It will be placed the day of the implant surgery and tighten to 25 N
  Interventions: Procedure: Citric acid abutment

INTERVENTIONS:
Procedure: Citric acid abutment — The implant surgery will be performed by 3rd year residents of the Postgraduate Program in Periodontology at UIC, supervised by a board-certified periodontist (J.V). Under local anaesthesia, a mid crestal incision will be performed and a full thickness flap will be raised. Implants will be placed following the manufacturer's recommendations. Implant shoulder (IS) will be placed 1 mm subcrestally, and a distance of ≥ 1.5 mm from adjacent natural tooth and ≥ 3 mm between implants will be always respected. Implant stability will be measured with Ostell ISQ. Straight definitive abutments (2 mm height) will be tightened to 25 N respecting the previous randomization procedure. One of the implants will receive an antibacterial- coated abutment (citric acid), while the other implant will receive a non-coated abutment (C). A protector cap will be screwed manually. Implant sites will be sutured with polypropylene 5/0 (Prolene Ethicon, USA) by simple stitches.

SUMMARY:
The use of dental implants is a predictable procedure to replace the missing tooth with high rates of success and survival. In addition, placing the abutment on the same day as the implant surgery is a safe and biologically sound procedure to minimize bone loss and peri-implant inflammation. Although citric acid antibacterial coating has never been tested in vivo, recent in vitro data support its clinical use due to its antibacterial effect at the abutment level.

This prospective randomized controlled clinical trial aims to evaluate the microbiological and inflammatory profile of implant abutments coated with citric acid.

DETAILED DESCRIPTION:
The study population will consist on patients referred to the Department of Periodontology at Universitat Internacional de Catalunya for the replacement of missing teeth and who meet the following inclusion criteria will be included consecutively in the study.

5.3.1. Inclusion criteria

* Patients with ≥18 years old.
* Systemically healthy patients.
* Patients with healthy periodontal status with a full mouth plaque index ≤ 20% (O'Leary, 1972) and full mouth bleeding index (Ainamo & Bay, 1975) before implant surgery.
* Need for at least one dental implant in maxillary and mandibular partially posterior edentulous healed sites.

5.3.2. Exclusion criteria

* Patients with some special conditions that could interfere surgical oral procedures.
* Patients with non-treated periodontal disease.
* Patients with uncontrolled systemic disease that could impair wound healing (i.e. Diabetes Mellitus).
* Pregnant women.
* Patients allergic to any metallic component of the materials.
* Need for bone or soft tissue reconstruction simultaneous to implant placement.
* Lack of primary stability during implant placement (i.e., insertion torque < 25 N, ISQ > 60)
* Smokers ≥ 10 cigarettes per day.
* Patients will be excluded from the study if they violate any of the criteria during the trial, as well as if they desire to withdraw the study or have any adverse reactions to the materials employed.

The primary outcome measure will be the reduction of biofilm formation at the test abutments compared with the control abutments at the 12 weeks 6 months, 1 year and 3 year of follow-up. Biofilm formation over abutments will be quantified with Ilumina sequencing analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥18 years old.
* Systemically healthy patients.
* Patients with healthy periodontal status with a full mouth plaque index ≤ 20% (O'Leary, 1972) and full mouth bleeding index (Ainamo & Bay, 1975) before implant surgery.
* Need for at least one dental implant in maxillary and mandibular partially posterior edentulous healed sites.

Exclusion Criteria:

* Patients with some special conditions that could interfere surgical oral procedures.
* Patients with non-treated periodontal disease.
* Patients with uncontrolled systemic disease that could impair wound healing (i.e. Diabetes Mellitus).
* Pregnant women.
* Patients allergic to any metallic component of the materials.
* Need for bone or soft tissue reconstruction simultaneous to implant placement.
* Lack of primary stability during implant placement (i.e., insertion torque < 25 N, ISQ > 60)
* Smokers ≥ 10 cigarettes per day.
* Patients will be excluded from the study if they violate any of the criteria during the trial, as well as those that desire to withdraw the study or have any adverse reactions to the materials employed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-03 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biofilm quantification | 12 weeks, 6 months, 1 and 3 years
  The primary outcome measure will be the reduction of biofilm formation at the test abutments compared with the control abutments at the 12 weeks, 6 months, 1 year and 3 years. Biofilm formation over the retrieved abutments will be quantified by means of Illumina sequencing analysis

SECONDARY OUTCOMES:
Protein expression markers | 12 weeks, 6 months, 1 and 3 years
  Quantification of protein expressions (IL-10 beta, IL-8 and TNF-beta) for the test and control abutments. This quantification will be performed at 12 weeks, 6 months, 1 and 3 years
Peri-implant disease incidence | 1 and 3 years
  The incidence of peri-implant disease will be assessed at 1 and 3 years attending to the 2017 World Workshop Classification

CONTACTS AND LOCATIONS:
Overall Officials: Javi Vilarrasa, Principal Investigator — Universitat Internacional de Catalunya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vilarrasa J, Pereira Couto C, Alvarez G, Carrio N, Gil J, Blanc V, Nart J. Microbiological, Inflammatory and Clinical Outcome of Citric Acid Passivated Definitive Abutments: Interim 12-Month Results From a Randomised Controlled Clinical Trial. J Clin Periodontol. 2025 Jun;52(6):813-825. doi: 10.1111/jcpe.14146. Epub 2025 Mar 11. PMID 40070156